CLINICAL TRIAL: NCT03781297
Title: Protocol for a Feasibility Study of Narrative Exposure Therapy in Homeless Individuals With Post-Traumatic Stress Disorder
Brief Title: Narrative Exposure Therapy Study for PTSD Among the Homeless Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Scientist, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017042
Record Dates: First submitted 2018-06-20; First posted 2018-12-19 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: PTSD
Keywords: Homeless Populations; PTSD; Narrative Exposure Therapy; Individual Therapy; Genealogy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: NET+G (Active Comparator): In addition to usual care, participants will receive six sessions of Narrative Exposure Therapy over six weeks plus the option to receive genealogical services.
  Interventions: Other: Narrative Exposure Therapy; Other: Genealogical Services
- Intervention: NET (Active Comparator): In addition to usual care, participants will receive six sessions of Narrative Exposure Therapy over six weeks.
  Interventions: Other: Narrative Exposure Therapy

INTERVENTIONS:
Other: Narrative Exposure Therapy — Narrative Exposure Therapy attempts to place the trauma within a narrative of the person's life. Anecdotal evidence of using this approach in the homeless population is that constructing an autobiography helps to give meaning to their problems and provide the initial steps in constructing a core sense of belonging and identity. Six sessions of individual therapy allows for participants to work with a therapist one-on-one to position their experiences of trauma within their life story.
Other: Genealogical Services — At the start of their involvement in the, study participants randomized to this group will be provided with the option to access services from a professional genealogist, to trace their family history. Participants will be made aware of the fact that new family information will be revealed through this process, and also be informed of the standard methods that will be used to extract this information which could involve research through publicly available historical records or voluntary DNA testing.
  Arms: Intervention: NET+G

SUMMARY:
The purpose of this study is to assess the acceptability and feasibility of delivering Narrative Exposure Therapy to homeless individuals with Post-Traumatic Stress Disorder.

In Ottawa, in 2015, there were 6,825 people using 500,191 bed nights in the city emergency shelters (Alliance to End Homelessness in Ottawa 2015 Annual Report) with approximately another 500 sleeping on the streets (The Homelessness Community Capacity Building Steering Committee 2008 Ottawa, ON). Mental health disorders, including substance abuse, are common in this population, are often under treated and can be a source of considerable distress and disability.

In addition to the high rates of mental disorder, there are three other significant factors which impact morbidity. First, a history of significant childhood trauma is common which impacts relationships and ability to cope with difficulties. It is increasingly recognized that a trauma informed approach to providing services to the homeless population is needed. There have been no randomized controlled trials of treatment of post-traumatic stress disorder in the homeless population. Second, brain dysfunction from head injuries and attention deficit disorder appear to be common. Problems with brain dysfunction can cause difficulties especially with attention, impulsivity and managing relationships. Finally, life for the marginally housed can be chaotic with day-to-day uncertainty over accommodation, income and security. This means that providing health services to this population requires a degree of flexibility in terms of who provides services, where and when.

These issues result in a population with complex needs that traditional mental health care is poorly equipped to serve. At present there is a clear gap in the provision of services that address the experience of trauma in homeless individuals. There are no services for trauma in publicly funded hospitals, which leaves private providers as the sole source of treatment. Other potential barriers include accounting for the effects of substance abuse, brain injury and "chaos" in this population. What the investigators are proposing is a pilot study to assess the feasibility and acceptability of providing a time-limited assessment and therapy (six sessions) within the shelter system to homeless individuals diagnosed with post-traumatic stress disorder.

DETAILED DESCRIPTION:
The purpose of this study is to assess the acceptability and feasibility of delivering Narrative Exposure Therapy to homeless individuals with Post-Traumatic Stress Disorder. This includes assessing the feasibility of recruiting sufficient numbers of participants, conducting a randomized trial in the shelter system and achieving adequate participant follow-up rates.

Study procedures will take place at shelters served by the Royal Ottawa Mental Health Centre's Psychiatric Outreach Team and Inner City Health, which are: The Shepherds of Good Hope, The Salvation Army, The Mission, Cornerstone Housing for Women, and other locations served by The Royal Ottawa's Psychiatric Outreach Team and Inner City Health.

Homeless individuals who meet criteria for PTSD will be offered, in addition to usual care, six sessions of Narrative Exposure Therapy either with or without the option of receiving services from a genealogist to supplement the process of exploring their life narrative. A total of 24 participants will be recruited into this study and will be randomized in a 1:1 allocation. At the start of their involvement in the study, participants randomized to receive genealogical services will be provided with the option to access services from a professional genealogist, to trace their family history. Participants will be made aware of the fact that new family information will be revealed through this process, and also be informed of the standard methods that will be used to extract this information which could involve research through publicly available historical records or voluntary DNA testing.

The primary outcomes for this study are acceptability - the investigators would deem the interventions acceptable if 50% of people approached consented to be randomized; and feasibility - the investigators would deem the study feasible if the planned sample size was recruited over a period of six months. Secondary outcomes include changes from baseline on relevant rating scales of symptoms, housing status, quality of life; and follow-up of participants three months from enrollment. This study will inform mental health treatment of this chronically underserved population.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* Be 18 years of age or older;
* Be referred to the study by the Psychiatric Outreach program at the Royal Ottawa Health Care Group or by Inner City Health;
* Meet DSM-5 criteria for post-traumatic stress disorder, as measured by the Mini International Neuropsychiatric Interview (MINI); and,
* Be homeless or vulnerably housed at the time of their screening visit, as measured by the Housing Status Questionnaire.

Exclusion Criteria:

Patients must not:

* Be unable to speak and understand English;
* Be unwilling to attend Narrative Therapy session for a period of six weeks;
* Be unwilling to return to a designated therapy location to complete study follow-up appointments;
* Be unwilling or unable to provide informed consent;
* Present to their study screening visit acutely intoxicated;
* Be, in the opinion of the Investigator, unlikely to commit to a 12-week study; or
* Pose a risk of harm to study staff or other clients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability measured by Recruitment Rates | 6 months
  The investigators would deem the interventions acceptable if 50% of people approached consented to participate in the study.
Feasibility measured by Sample Size | 6 months
  The investigators would deem a larger study to be feasible if the investigators could identify the planned sample size (n=24) over a six month period.

SECONDARY OUTCOMES:
Acceptability & Feasibility of Collecting Outcome Data measured by Retention Rates | 6 months
  Collecting outcome data within this population will be determined acceptable/feasible if dropout and incomplete outcome assessment is limited to 25% of participants three months after the intervention.
Change in Post-Traumatic Stress Disorder (PTSD) symptoms as measured by the PTSD Checklist for DSM-5 (PCL-5) | Baseline, Week 8, Week 12
  The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. The PCL-5 will be collected as part of the Narrative Exposure Therapy Session to quantify PTSD symptoms and traumatic experiences. Blevins et al. (2015) demonstrated that PCL-5 scores exhibited strong internal consistency (α = .94), test-retest reliability (r = .82), and convergent (rs = .74 to .85) and discriminant (rs = .31 to .60) validity.
Change in Housing Status as measured by Self-Report from Participants | Baseline, Week 4, Week 8, Week 12
  Any changes in housing status during the study period (including follow-up period) will be noted. This will be assessed by asking the participants directly about their current housing status throughout the study period.
Change in scores on Health-Related Quality of Life and Functioning as measured by the 20-item Medical Outcomes Survey Short Form Health Survey (SF-20) | Baseline, Week 4, Week 8, Week 12
  This is a 20-item questionnaire that assesses various health outcomes, and the extent to which health related problems interfere with daily life. The SF-20 [27] uses questions related to 8 domains: physical functioning, role functioning (physical), bodily pain, general health, vitality, social functioning, role functioning (emotional) and mental health. Each item is scored on a scale of 0 to 100 and then averaged to obtain a sub-scale score. Sub-scale scores on the SF-20 are rated on a scale from 0 to 100, with high scores indicating a higher degree of functionality.
Change in Scores for Substance Use/Misuse as measured by the Addiction Severity Index (ASI) | Baseline, Week 4, Week 8, Week 12
  A semi-structured interview used to assess severity of substance abuse problems. Questions are related to the following seven potential areas that could be impacted by substance use: Medical, Employment/Support Status, Legal, Family/Social and Psychiatric, as well as Alcohol specific and Drug specific questions. This interview gathers information on current (past 30 days) and lifetime substance abuse.
  Severity ratings are based on the following 10 point scale (0-9): 0-1 No real problem, treatment not indicated; 2-3 Slight problem, treatment probably not necessary; 4-5 Moderate problem, some treatment indicated; 6-7 Considerable problem, treatment necessary; 8-9 Extreme problem, treatment absolutely necessary.
Change in Scores for Alcohol Use/Misuse as measured by the Alcohol Use Disorder Identification Test (AUDIT) | Baseline, Week 4, Week 8, Week 12
  The AUDIT questionnaire is designed to assess the following four dimensions of alcohol misuse: Alcohol consumption (3 items); Drinking behaviour (3 items); Adverse reactions (2 items); Alcohol-related problems (2 items).
  The first three items of the AUDIT (AUDIT-C) will be used as a screening questionnaire. Participants who score above 4 on the first three items of the AUDIT-C will be asked to complete the Full AUDIT. In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
  For the Full AUDIT, a score of (0-7) indicates low-risk. (8-15) indicates risky or a hazardous level of drinking behaviours. (16-19) indicates high-risk or a harmful level of drinking behaviours. A score of (20 or more) indicates high risk alcohol related behaviours and an almost certainty of dependence.
Change in Health Care Costs as measured by Self-Report Questionnaire | Baseline, Week 4, Week 8, Week 12
  A questionnaire has been created by the research team to capture data related to health care costs. The Health Care Costs questionnaire is an 11-item questionnaire that evaluates the effect of mental health on an individual's ability to work and perform regular activities.
  Specifically, elements from the Client Service Receipt Inventory (CSRI) and the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI: SHP) as well as other health cost indicators used in previous studies conducted by the Principal Investigator.

OTHER OUTCOMES:
Severity of Attention Deficit Hyperactivity Disorder (ADHD) as measured by the ADHD Self-Report Scale (ASRS) | Baseline
  The ASRS an 18-item self-report questionnaire that assesses the inattentive (6 items) and hyperactive/impulsive (12 items) dimensions of ADHD. Participants are asked to rate items of a five-point Likert scale from "Never" (0) to "Very Often" (4), with total scores on each sub-scale ranging from 0-24 (inattentive) and 0-48 (hyperactive/impulsive). Scores between (0-16) indicate an unlikely presentation of ADHD. Scores between (17-23) indicate a likely presentation of ADHD. Scores of (24) or greater indicate a highly likely presentation of ADHD.
Level of Cognitive Functioning as measured by the Montreal Cognitive Assessment (MoCA) | Baseline
  Cognitive functioning will be assessed using the Montreal Cognitive Assessment (MoCA), which can be administered in ten minutes and includes the assessment of the following cognitive skills: alternating trail making; visuocontructional skills (cube); visuocontructional skills (clock); naming; memory; attention; sentence repetition; verbal fluency; abstraction; delayed recall; and, orientation [33]. Total possible scores for the MoCA range from 0 to 30, with a score of 26 or above being considered normative. This measure will be used in the initial assessment only for the purposes of tailoring the intervention for the individual.
Diagnosis of PTSD as measured by the MINI International Neurpsychiatric Interview | Baseline
  A clinical interview with a delegated study staff member will be conducted with each participant enrolled in the study. This interview will be guided by the Mini International Neurpsychiatric Interview (MINI) to confirm a diagnosis of PTSD.
Demographic Characteristics as measured by Self-Report | Baseline
  Includes assessments of gender identity, age, marital status, ethnicity, primary language, level of education, Canadian Armed Forces membership and sexual identity

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatcher, MD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Fazel S, Khosla V, Doll H, Geddes J. The prevalence of mental disorders among the homeless in western countries: systematic review and meta-regression analysis. PLoS Med. 2008 Dec 2;5(12):e225. doi: 10.1371/journal.pmed.0050225. PMID 19053169
- [Background] Fazel S, Geddes JR, Kushel M. The health of homeless people in high-income countries: descriptive epidemiology, health consequences, and clinical and policy recommendations. Lancet. 2014 Oct 25;384(9953):1529-40. doi: 10.1016/S0140-6736(14)61132-6. PMID 25390578
- [Background] Torchalla I, Strehlau V, Li K, Aube Linden I, Noel F, Krausz M. Posttraumatic stress disorder and substance use disorder comorbidity in homeless adults: Prevalence, correlates, and sex differences. Psychol Addict Behav. 2014 Jun;28(2):443-52. doi: 10.1037/a0033674. Epub 2013 Aug 5. PMID 23915373
- [Background] Kumar SA, Brand BL, Courtois CA. The need for trauma training: Clinicians' reactions to training on complex trauma. Psychol Trauma. 2022 Nov;14(8):1387-1394. doi: 10.1037/tra0000515. Epub 2019 Oct 3. PMID 31580137
- [Background] Litz BT, Stein N, Delaney E, Lebowitz L, Nash WP, Silva C, Maguen S. Moral injury and moral repair in war veterans: a preliminary model and intervention strategy. Clin Psychol Rev. 2009 Dec;29(8):695-706. doi: 10.1016/j.cpr.2009.07.003. Epub 2009 Jul 29. PMID 19683376
- [Background] Dinnen S, Kane V, Cook JM. Trauma-informed care: a paradigm shift needed for services with homeless veterans. Prof Case Manag. 2014 Jul-Aug;19(4):161-70; quiz 171-2. doi: 10.1097/NCM.0000000000000038. PMID 24871433
- [Background] Hopper E, Bassuk E, Olivet J. Shelter from the storm: Trauma-informed care in homelessness service settings. The Open Health Services and Policy Journal 2010; 3: 80-100.
- [Background] Topolovec-Vranic J, Ennis N, Colantonio A, Cusimano MD, Hwang SW, Kontos P, Ouchterlony D, Stergiopoulos V. Traumatic brain injury among people who are homeless: a systematic review. BMC Public Health. 2012 Dec 8;12:1059. doi: 10.1186/1471-2458-12-1059. PMID 23216886
- [Background] To MJ, O'Brien K, Palepu A, Hubley AM, Farrell S, Aubry T, Gogosis E, Muckle W, Hwang SW. Healthcare Utilization, Legal Incidents, and Victimization Following Traumatic Brain Injury in Homeless and Vulnerably Housed Individuals: A Prospective Cohort Study. J Head Trauma Rehabil. 2015 Jul-Aug;30(4):270-6. doi: 10.1097/HTR.0000000000000044. PMID 24651000
- [Background] Salavera C, Antonanzas JL, Bustamante JC, Carron J, Usan P, Teruel P, Bericat C, Monteagudo L, Larrosa S, Tricas JM, Lucha O, Noe R, Jarie L, Cerra R. Comorbidity of attention deficit hyperactivity disorder with personality disorders in homeless people. BMC Res Notes. 2014 Dec 16;7:916. doi: 10.1186/1756-0500-7-916. PMID 25516377
- [Background] Farrell SJ, Huff J, MacDonald SA, Middlebro A, Walsh S. Taking it to the street: a psychiatric outreach service in Canada. Community Ment Health J. 2005 Dec;41(6):737-46. doi: 10.1007/s10597-005-6430-7. PMID 16328586
- [Background] Schauer M, Neuner F, Elbert T. Narrative Exposure Therapy: A short term treatment for traumatic stress disorders. 2nd ed. Cambridge, MA: Hogrefe Publishing; 2011.
- [Background] Cloitre M. Effective psychotherapies for posttraumatic stress disorder: a review and critique. CNS Spectr. 2009 Jan;14(1 Suppl 1):32-43. PMID 19169192
- [Background] Morkved N, Hartmann K, Aarsheim LM, Holen D, Milde AM, Bomyea J, Thorp SR. A comparison of Narrative Exposure Therapy and Prolonged Exposure therapy for PTSD. Clin Psychol Rev. 2014 Aug;34(6):453-67. doi: 10.1016/j.cpr.2014.06.005. Epub 2014 Jun 26. PMID 25047447
- [Background] van Minnen A, Arntz A, Keijsers GP. Prolonged exposure in patients with chronic PTSD: predictors of treatment outcome and dropout. Behav Res Ther. 2002 Apr;40(4):439-57. doi: 10.1016/s0005-7967(01)00024-9. PMID 12002900
- [Background] Monson CM, Schnurr PP, Resick PA, Friedman MJ, Young-Xu Y, Stevens SP. Cognitive processing therapy for veterans with military-related posttraumatic stress disorder. J Consult Clin Psychol. 2006 Oct;74(5):898-907. doi: 10.1037/0022-006X.74.5.898. PMID 17032094
- [Background] Zang Y, Hunt N, Cox T. A randomised controlled pilot study: the effectiveness of narrative exposure therapy with adult survivors of the Sichuan earthquake. BMC Psychiatry. 2013 Jan 31;13:41. doi: 10.1186/1471-244X-13-41. PMID 23363689
- [Background] Hatcher S, Coupe N, Wikiriwhi K, Durie SM, Pillai A. Te Ira Tangata: a Zelen randomised controlled trial of a culturally informed treatment compared to treatment as usual in Maori who present to hospital after self-harm. Soc Psychiatry Psychiatr Epidemiol. 2016 Jun;51(6):885-94. doi: 10.1007/s00127-016-1194-7. Epub 2016 Mar 8. PMID 26956679
- [Background] Henry, M., Cortes, A., Shivji, A., & Buck, K. (2014). Part 1: point-in-time estimates of homelessness. In The Annual Homeless Assessment Report to Congress 2014 (pp. 1-62).
- [Background] Gaetz, S., Gulliver, T., & Richter, T. (2014). The state of homelessness in Canada 2014. Canadian Homelessness Research Network.
- [Background] Thompson AE, Anisimowicz Y, Miedema B, Hogg W, Wodchis WP, Aubrey-Bassler K. The influence of gender and other patient characteristics on health care-seeking behaviour: a QUALICOPC study. BMC Fam Pract. 2016 Mar 31;17:38. doi: 10.1186/s12875-016-0440-0. PMID 27036116
- [Background] Luoma JB, Martin CE, Pearson JL. Contact with mental health and primary care providers before suicide: a review of the evidence. Am J Psychiatry. 2002 Jun;159(6):909-16. doi: 10.1176/appi.ajp.159.6.909. PMID 12042175
- [Background] O'toole TP, Conde-Martel A, Gibbon JL, Hanusa BH, Freyder PJ, Fine MJ. Substance-abusing urban homeless in the late 1990s: how do they differ from non-substance-abusing homeless persons? J Urban Health. 2004 Dec;81(4):606-17. doi: 10.1093/jurban/jth144. PMID 15466842
- [Background] Lev-Ran S, Le Strat Y, Imtiaz S, Rehm J, Le Foll B. Gender differences in prevalence of substance use disorders among individuals with lifetime exposure to substances: results from a large representative sample. Am J Addict. 2013 Jan;22(1):7-13. doi: 10.1111/j.1521-0391.2013.00321.x. PMID 23398220
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Carver DJ, Chapman CA, Thomas VS, Stadnyk KJ, Rockwood K. Validity and reliability of the Medical Outcomes Study Short Form-20 questionnaire as a measure of quality of life in elderly people living at home. Age Ageing. 1999 Mar;28(2):169-74. doi: 10.1093/ageing/28.2.169. PMID 10350414
- [Background] McLellan AT, Luborsky L, Woody GE, O'Brien CP. An improved diagnostic evaluation instrument for substance abuse patients. The Addiction Severity Index. J Nerv Ment Dis. 1980 Jan;168(1):26-33. doi: 10.1097/00005053-198001000-00006. PMID 7351540
- [Background] Zanis DA, McLellan AT, Cnaan RA, Randall M. Reliability and validity of the Addiction Severity Index with a homeless sample. J Subst Abuse Treat. 1994 Nov-Dec;11(6):541-8. doi: 10.1016/0740-5472(94)90005-1. PMID 7884837
- [Background] Carey KB, Carey MP, Chandra PS. Psychometric evaluation of the alcohol use disorders identification test and short drug abuse screening test with psychiatric patients in India. J Clin Psychiatry. 2003 Jul;64(7):767-74. doi: 10.4088/jcp.v64n0705. PMID 12934976
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Adler LA, Spencer T, Faraone SV, Kessler RC, Howes MJ, Biederman J, Secnik K. Validity of pilot Adult ADHD Self- Report Scale (ASRS) to Rate Adult ADHD symptoms. Ann Clin Psychiatry. 2006 Jul-Sep;18(3):145-8. doi: 10.1080/10401230600801077. PMID 16923651
- [Background] Rossetti HC, Lacritz LH, Cullum CM, Weiner MF. Normative data for the Montreal Cognitive Assessment (MoCA) in a population-based sample. Neurology. 2011 Sep 27;77(13):1272-5. doi: 10.1212/WNL.0b013e318230208a. Epub 2011 Sep 14. PMID 21917776
- [Background] Cocks K, Torgerson DJ. Sample size calculations for pilot randomized trials: a confidence interval approach. J Clin Epidemiol. 2013 Feb;66(2):197-201. doi: 10.1016/j.jclinepi.2012.09.002. Epub 2012 Nov 27. PMID 23195919
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics 2005; 4: 287-91.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Derived] Edgar NE, Bennett A, Dunn NS, MacLean SE, Hatcher S. Feasibility and acceptability of Narrative Exposure Therapy to treat individuals with PTSD who are homeless or vulnerably housed: a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Apr 15;8(1):83. doi: 10.1186/s40814-022-01043-x. PMID 35428344